CLINICAL TRIAL: NCT02908113
Title: Sensory Maturation of Preterm Infants: From Visual Sensitivity to Multisensory Perception
Brief Title: Visual Perception in Preterm Infants
Acronym: PREMAVISION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6123
Record Dates: First submitted 2016-08-26; First posted 2016-09-20 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2016-10

CONDITIONS: Pediatrics
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preterm infants (Other): physiological data collection, behavioral, cerebral hemodynamics, physical environmental newborns studied in response to visual stimuli / auditory or visual-auditory calibrated
  Interventions: Behavioral: collection data; Behavioral: IRM
- term infants (Other): physiological data collection, behavioral, cerebral hemodynamics, physical environmental newborns studied in response to visual stimuli / auditory or visual-auditory calibrated
  Interventions: Behavioral: collection data; Behavioral: IRM

INTERVENTIONS:
Behavioral: collection data
Behavioral: IRM

SUMMARY:
We aim to increase our knowledge of the impact of preterm birth on the maturation of the visual and auditory systems and on the development of multisensory perception

Specifically, we aim to evaluate the preterm infants' capabilities of detection and discrimination of different visual and auditory stimuli according to gestational age, post menstrual age and the duration of the postnatal life.

A secondary aim is to compare this competencies in preterm and full term control art term equivalent age.

The final aim is to optimize the hospital environment in order to make it correspond to the expectations and sensory abilities of very preterm infants.

Our hypothesis is that preterm birth exposes the infants to numerous atypical stimuli which could accelerate the processes of sensory maturation

ELIGIBILITY:
Inclusion Criteria:

* Newborn less than 32 weeks PMA hospitalized in the Hospital of Hautepierre, Strasbourg, France)
* Consent obtained from both parents
* Social insurance coverage

Exclusion Criteria:

* Any known malformation
* Brain lesions discovered on brain ultrasound (Intra-Ventricular hemorrhage grade III or IV periventricular Leukomalacia).
* Unstable clinical State
* Retinopathy Of Prematurity stage> 2 or in zone 1
* Family history of abnormal color vision.
* Abnormalities in auditory testing
* Transfer to another hospital expected before 40 week PMA

Ages: 23 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
visual stimulus detection with luminance | 3 months
  in "green" condition in hospital, luminance ( 100 and 300 lux ) and color (blue- red-yellow- white) variables
auditory stimulus detection with parents voice | 3 months
  use parents voice, pure sound of 500 Hz

SECONDARY OUTCOMES:
behavioral responsiveness to visual stimuli calibrated collected from video recordings | 3 months
  Evaluate the facial expression of the imitation abilities in preterm and term neonates at term. The interpretation of the behavioral responses of newborns to mimic presented by the experimenter will be working independently by two observers with a coding grid

CONTACTS AND LOCATIONS:
Overall Officials: Claire KOENIG ZORES, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôiptaux Universitaires, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No